CLINICAL TRIAL: NCT00038090
Title: Thalidomide-Dexamethasone for Multiple Myeloma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-070
Record Dates: First submitted 2002-05-28; First posted 2002-05-29 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Thalidomide; Thalomid; Dexamethasone; Decadron
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Thalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thalidomide + Dexamethasone (Experimental)
  Interventions: Drug: Thalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Thalidomide — 100 mg capsules by mouth daily each evening
  Other Names: Thalomid
Drug: Dexamethasone — 20 mg/m^2 taken by mouth each morning on days 1-4, 9-12 and 17-20.
  Other Names: Decadron

SUMMARY:
Objective is to assess the activity of the combination of thalidomide and dexamethasone in patients with previously untreated multiple myeloma.

DETAILED DESCRIPTION:
This study will examine the potential efficacy of thalidomide-dexamethasone in the treatment of patients with previously untreated multiple myeloma.

* Thalidomide is supplied as 50 mg capsules to be taken by mouth.
* Thalidomide 200 mg daily each evening at bedtime increasing by 100-200 mg increments (according to patient tolerability) every 4 weeks.

For elderly patients, or those with poor performance status or comorbid conditions which may affect tolerance of the thalidomide-dexamethasone combination, the initial dose may be reduced by 50-100 mg decrements and escalated weekly by 50-100 mg increments to tolerance. For patients who experience significant toxicity (> grade 2) or are otherwise unable to tolerate this drug combination, the dose will be reduced by 50-100 mg decrements. For some patients with > grade 2 toxicity, it may be necessary to hold the thalidomide dose until improvement of the side effect with subsequent resumption of the dose after dose reduction as outlined above.

Dexamethasone 20mg/m2 each morning after breakfast on days 1-4, 9-12, 17-20, with a repeat cycle after a 1-2 week rest period. In case of partial remission, maintenance treatment with thalidomide alone will be continued for as long as remission is sustained at a dose free of side effects.

For patients achieving CR, consolidation with thalidomide-dexamethasone for 4-6 months followed by follow-up without maintenance treatment. No maximum trial period is planned.

At relapse patients may be reinitiated on the original thalidomide-pulse dexamethasone program and responding patients may be maintained on thalidomide alone (CR) or daily thalidomide and dexamethasone (days 1-4) until relapse.

Patients who experience significant toxicity (grade 2 or more) at any time during therapy will receive a lower dose after treatment is interrupted.

In an attempt to avoid deep venous thrombosis, all patients for whom anticoagulation is not contraindicated will be offered therapeutic anticoagulation (INR 1.5-2.5) with coumadin or therapeutic doses of low molecular weight heparin.

Patients must be willing to return for evaluation every 4 weeks since thalidomide may only be prescribed for 28 day intervals.

ELIGIBILITY:
* Previously untreated patients with symptomatic or progressive asymptomatic multiple myeloma. Criteria for progression among patients with asymptomatic disease include new lytic bone lesions, rise of serum myeloma protein to >5.0 gm/dl or fall of Hgb to <10.5 gm/dl.
* Overt infection or unexplained fever should be resolved before treatment or treated concurrently with antibiotics.
* Patients must provide written informed consent indicating that they are aware of the investigational nature of this study.
* Patients with idiopathic monoclonal gammopathy or stable asymptomatic myeloma are ineligible.
* Patients whose only prior therapy has been with local radiotherapy or alpha interferon are eligible.
* Patients treated with steroids in order to stabilize disease within 60 days prior to enrollment are eligible.
* Patients exposed to longer periods of high-dose glucocorticoid, or with any exposure to thalidomide or alkylating agent are ineligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2000-06; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Response Rate | Baseline, with each course and monthly tests

CONTACTS AND LOCATIONS:
Overall Officials: Donna M Weber, M.D., Study Chair — UT MD Anderson Cancer Center
Locations (1):
- University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org